CLINICAL TRIAL: NCT02680067
Title: Near InfraRed Fluorescence Imaging of Lymphatic Transport Using Indocyanine Green
Brief Title: NIR Fluorescence Imaging of Lymphatic Transport Using ICG
Acronym: NIR-ICG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine, Chief of Allergy, Immunology & Rheumatology Division, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSRB 54038; R01AR056702 (NIH)
Record Dates: First submitted 2015-12-07; First posted 2016-02-11 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Healthy Individual; Lymphatic Transport; Near InfraRed; Imaging; Indocyanine Green; ICG; NIR; NIR-ICG; MSImager; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Healthy individuals and subjects that have rheumatoid arthritis may participate in the developmental arm. Healthy individuals may participate in the clearance arm. There will be no randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Developmental arm - Healthy or rheumatoid arthritis subjects (Experimental): Subjects in the developmental arm will have a minimum of two study visits to determine the optimal conditions for visualizing lymphatic transport in the upper extremities. Concentrations of 0.1 mg/ml of Indocyanine Green (ICG) will be injected intradermally into the web spaces of the hands in both upper extremities. Multispectral video and still images will be recorded using the MultiSpectral Imaging System (MSImager). An ultrasound of the upper extremities may be performed after the ICG fluorescence is observed. The exam will help identify the location of the lymphatic vessels and nodes in the areas fluoresced.
  Interventions: Drug: Indocyanine Green; Device: MultiSpectral Imaging System
- Clearance arm - Healthy individuals (Experimental): Subjects in the clearance arm will have an initial study visit that involves injections of 0.1 mg/ml of Indocyanine Green (ICG) intradermally into the web spaces of the hands in both upper extremities. Multispectral video and still images will be recorded using the MultiSpectral Imaging System (MSImager). Follow up imaging sessions will occur weekly for three weeks for a minimum of four study visits total.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — A trained physician will inject 0.1 ml of Indocyanine Green into the web spaces of the hands in both upper extremities. Subjects may have up to five study visits to confirm feasibility, safety, and reproducibility.
  Other Names: ICG; IC-Green; 17478-701-02
Device: MultiSpectral Imaging System — Once the Indocyanine Green is injected, the contrast is expected to fluoresce underneath the MultiSpectral Imaging System. Multispectral video and still images will be recorded at the study visits.
  Other Names: MSImager
  Arms: Developmental arm - Healthy or rheumatoid arthritis subjects

SUMMARY:
In this phase 1 study, the lymphatic transport will be examined using Near InfraRed Indocyanine Green fluorescence imaging (NIR-ICG) of the upper extremities in healthy individuals using a MultiSpectral Imaging System (MSImager).

DETAILED DESCRIPTION:
Lymphedema from various etiologies (i.e. infection, cancer, surgery, and rheumatoid arthritis) remains a major health concern. Efforts to develop effective treatments for this condition have been limited by the absence of quantitative outcome measures for lymphatic function. Published articles have supported the fact that human lymphatic contractions can be readily visualized after intradermal administration of micrograms of Indocyanine Green using laser-induced fluorescence. The use of lasers imposes a risk of eye injury that requires protective eyewear. To address the risk of laser-induced injury, an imaging system was developed by Drs. Ronald Wood and Jay Reeder in a collaborative effort at the University of Rochester. In place of a laser, this system utilizes a tungsten-halogen lamp fitted with a bandpass filter and a multispectral camera for real-time image acquisition and display. This phase 1 study will examine the validity and reliability of this instrument to measure lymphatic transport, contractions, and pressure in the arms of healthy research subjects and establish baseline parameters for subsequent evaluation of rheumatoid arthritis patients in later studies. Indocyanine Green is a dye that has been used clinically for over 50 years to evaluate hepatic clearance, cardiovascular function testing, and retinal angiography. Indocyanine Green has typically been administered intravenously at concentrations of 2.5 mg/ml at total doses of 25 mg in adults. In this study, intradermal administration of micrograms of Indocyanine Green will be used to establish useful dose ranges and concentrations. The dosage regimen for this study is based on prior demonstrations in published articles of successful noninvasive imaging of lymphatic contractions after intradermal administration of microgram amounts of Indocyanine Green.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Subjects can be either gender but must be at least 18 years old.
* Rheumatoid arthritis subjects may fulfill 2010 American College of Rheumatology criteria.
* Active rheumatoid arthritis subjects, with at least 2 tender or swollen joints.
* Subjects participating in the clearance arm of the study must not have ICG injections for at least 10 weeks.

Exclusion Criteria:

* Individuals with active systemic disorders or inflammatory conditions other than rheumatoid arthritis, (such as chronic infections with hepatitis B, hepatitis C or HIV) that would confound the study results.
* Known sensitivity to iodine because of residual iodide in Indocyanine Green
* Pregnant women should not participate.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Contraction Rate | 36 months
  The contraction rate is measured as lymphatic vessel contractions/min in the dominant lymphatic vessel efferent to the injection site using the MultiSpectral Imaging System (MSImager) that captures real time movies. The MSImager software analyses the signal intensity to determine the contraction rate.

SECONDARY OUTCOMES:
Lymphatic Pressure | 36 months
  The lymphatic pressure is measured using a transparent cuff and the Multispectral Imaging System to determine indirect lymphatic pressure and recorded as mm Hg.

OTHER OUTCOMES:
Clearance | 36 months
  The change in Indocyanine Green signal intensity (arbitrary units) over time is measured by observing the fluorescence using the Multispectral Imaging System. The MSImager software analyses the signal intensity.
Lymphatic Speed | 36 months
  Speed with which an Indocyanine Green bolus moves through a lymphatic vessel recorded as mm -sec-1 using the Multispectral Imaging System. The MSImager software analyses the signal speed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD/MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information of any type may be shared with researchers at other institutions. Subjects will be made aware of this in the informed consent form.

REFERENCES:
- [Derived] Rahimi H, Bell R, Bouta EM, Wood RW, Xing L, Ritchlin CT, Schwarz EM. Lymphatic imaging to assess rheumatoid flare: mechanistic insights and biomarker potential. Arthritis Res Ther. 2016 Sep 1;18:194. doi: 10.1186/s13075-016-1092-0. PMID 27586634
- See also: Allergy, Immunology, and Rheumatology Clinical Trials — https://www.urmc.rochester.edu/medicine/allergy/patients-families/clinical-trials.aspx
- Available data/document: Arthritis Research & Therapy Publication — http://arthritis-research.biomedcentral.com/articles/10.1186/s13075-016-1092-0 — Lymphatic imaging to assess rheumatoid flare: mechanistic insights and biomarker potential.